CLINICAL TRIAL: NCT04180215
Title: A Phase I/II Study of TheraT® Vector(s) Expressing Human Papillomavirus 16 Positive (HPV 16+) Specific Antigens in Patients With HPV 16+ Confirmed Cancers
Brief Title: A Phase 1/2 Study in Patients With HPV16+ Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma and Other Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hookipa Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-200-001; 2019-000907-34 (EudraCT Number)
Record Dates: First submitted 2019-09-20; First posted 2019-11-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: HPV-Related Squamous Cell Carcinoma
Keywords: Vaccine; Gene Therapy; TheraT®; E7E6; HPV 16 E7E6; HNSCC; HPV 16+ head and neck squamous cell cancer; Oropharyngeal cancer; HPV16; HPV 16; Head and neck cancer; Carcinoma; Carcinoma, squamous cell; Squamous cell carcinoma of head and neck; Neoplasms, squamous cell; Head and neck neoplasms; Pembrolizumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Head and Neck Neoplasms; Carcinoma; Carcinoma, Squamous Cell; Neoplasms, Squamous Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Ph I, Group 1 and Group 2 (Experimental): Patients with HPV 16+ HNSCC or Non-HNSCC who had tumor progression or recurrence on standard of care therapy.
  Interventions: Drug: HB-201 intravenous administration.
- Ph I, Group 3 and Group 4 (Experimental): Patients with HPV 16+ HNSCC or Non-HNSCC who had tumor progression or recurrence on standard of care therapy.
  Interventions: Drug: HB-202 intravenous administration alternating with HB-201 intravenous administration.
- Ph II, Group B (Experimental): Patients with HPV 16+ HNSCC who are eligible to receive immune checkpoint inhibitor as part of standard of care.
  Interventions: Drug: HB-201 intravenous administration + standard of care regimen including pembrolizumab.
- Ph II, Group E (Experimental): Patients with HPV 16+ HNSCC who are eligible to receive pembrolizumab as part of 1L standard of care.
  Interventions: Drug: HB-202 / HB-201 alternating intravenous administration + standard of care regimen including pembrolizumab.
- Ph II, Group F (Experimental): Patients with HPV 16+ cancers who had tumor progression or recurrence on standard of care therapy and who are eligible to receive pembrolizumab as part of 2L+ standard of care..
  Interventions: Drug: HB-202 / HB-201 alternating intravenous administration + pembrolizumab.
- Ph I, sub-study (Experimental): Patients with HPV 16+ HNSCC who had tumor progression or recurrence on standard of care therapy
  Interventions: Drug: HB-201 or HB-201/HB-202 alternating treatment using CD8 PET Tracer (Zr-Df-IAB22M2C)

INTERVENTIONS:
Drug: HB-201 intravenous administration. — Dose / Schedule determined by 3+3 dose escalation (3 to 6 patients per cohort).
  Arms: Ph I, Group 1 and Group 2
Drug: HB-202 intravenous administration alternating with HB-201 intravenous administration. — Dose / Schedule determined by 3+3 dose escalation (3 to 6 patients per cohort).
  Arms: Ph I, Group 3 and Group 4
Drug: HB-201 intravenous administration + standard of care regimen including pembrolizumab. — Dose Expansion
  Arms: Ph II, Group B
Drug: HB-202 / HB-201 alternating intravenous administration + pembrolizumab. — Dose Expansion
  Arms: Ph II, Group F
Drug: HB-202 / HB-201 alternating intravenous administration + standard of care regimen including pembrolizumab. — Dose Expansion
  Arms: Ph II, Group E
Drug: HB-201 or HB-201/HB-202 alternating treatment using CD8 PET Tracer (Zr-Df-IAB22M2C) — Dose escalation; 10 patients
  Arms: Ph I, sub-study

SUMMARY:
This is a First in Human (FIH) Phase I/II, multinational, multicenter, open-label study of HB-201 single vector therapy and HB-201 & HB-202 two-vector therapy in patients with HPV 16+ confirmed cancers comprising two parts: Phase I Dose Escalation and Phase II Dose Expansion.

DETAILED DESCRIPTION:
HB-201 and HB-202 are study drugs which are designed to train the body to recognize and fight substances found in HPV 16+ cancer. This trial studies the safety and anti-cancer effect of HB-201 and HB-202 in people.

The trial is enrolling patients with metastatic/recurrent head and neck cancer who have not yet received treatment in this setting (1L, first line) and who are eligible to receive pembrolizumab as part of their standard of care. This trial is also enrolling patients with metastatic/recurrent head and neck who have received prior treatment in this setting (2L+, second and later line) who are eligible to receive pembrolizumab as part of their standard of care. Patients will receive the study drugs in addition to their pembrolizumab standard of care regimen.

ELIGIBILITY:
Inclusion Criteria

All Patients:

* Documentation of confirmed HPV 16+ cancer via genotype testing.
* ≥ 1 measurable lesion by imaging for tumor response following RECIST
* ECOG performance status of 0 to 1.
* Prior curative radiation therapy and prior focal palliative completed per protocol-specified wash-out windows.
* Screening laboratory values must meet protocol-specified criteria.
* Able to provide tumor tissue following last treatment, unless otherwise agreed.

Treatment Group E or Group F:

* Documentation of confirmed head and neck squamous cell carcinoma.
* Eligible to receive pembrolizumab, per standard of care and product label.
* Group E: this group includes first line / 1L patients who have not yet received treatment in the metastatic/recurrent setting.
* Group F: Tumor progression or recurrence on standard of care therapy, including ≥1 systemic therapy.

Imaging Sub-Study (for specific participants at Memorial Sloan Kettering Cancer Center only):

* Meeting requirements of inclusion criteria for Treatment Group 1 or Group 3.
* At least 1 non-irradiated measurable lesion documented through imaging.

Exclusion Criteria:

All patients:

* Metastatic central nervous system disease, and/or carcinomatous meningitis.
* Any serious or uncontrolled medical disorder that, in the opinion of the Investigator, may increase the risk associated with study participation / treatment administration.
* Concurrent malignancy that is clinically significant or requires active intervention, unless protocol-defined criteria are met.
* Active, known or suspected, autoimmune or inflammatory disorders requiring immunosuppressive therapy.
* Has a life expectancy of less than 3 months.
* Any toxicities attributed to systemic prior anticancer therapy o that have not resolved to Grade 1 or baseline prior to the first administration of study drug, unless protocol-defined criteria is met.
* Not meeting the protocol-specified washout periods for prohibited medications.
* Prior anaphylactic reaction to or known allergy or hypersensitivity to investigational product(s) or any of the excipients of the investigational product(s).
* Positive hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody, indicating acute or chronic infection.
* Known history of acquired immunodeficiency syndrome.

For patients in Groups E or F and certain backfill cohorts:

* History of severe hypersensitivity reaction to or other contraindication to receiving pembrolizumab.
* History of/Presently having non-infectious pneumonitis requiring treatment.
* Was discontinued due to a Grade 3 or higher immune-related AE (irAE) after receiving prior therapy with check point inhibitors.

Imaging Sub-Study (for specific participants at Memorial Sloan Kettering Cancer Center only):

* Having splenic disorders or prior splenectomy, and can compromise protocol objectives per Investigator and/or Sponsor.
* Meeting requirements of exclusion criteria for Treatment Group 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Phase I Dose Escalation: Determine Phase II dose based on incidence of dose-limiting toxicities. | From dosing until 21-28 days after first dose
  Determine the recommended Phase II dose in terms of safety and tolerability for intravenously administered HB-201, and intravenously administered HB-202 by assessing drug limiting toxicities.
Phase II Dose Expansion: Number of participants with preliminary antitumor activity based on objective response rate. | Until progression, (estimated up to 30-months)
  Assess the preliminary antitumor activity of dosage regimens of HB-201 and HB-202 using Response Evaluation Criteria in Solid Tumors (RECIST) to determine objective response rate (ORR).

SECONDARY OUTCOMES:
Phase I Dose Escalation: Number of participants with adverse events (type, frequency, severity). | From informed consent through 30 days after last dose.
  Assess the safety and tolerability of dosage regimens of HB-201 and HB-202 by monitoring the type, frequency, and severity of AEs and SAEs by monitoring the type, frequency, and severity of AEs and SAEs.
Phase I Dose Escalation: Number of participants with preliminary antitumor activity based on objective response rate and disease control rate. | Until progression, (estimated up to 30-months)
  Assess the preliminary antitumor activity of dosage regimens of HB-201 and HB-202 using RECIST and iRECIST
Phase II Dose Expansion: Number of participants with confirmed duration of preliminary antitumor activity. | Up to 30-months (until progression)
  Confirm duration of preliminary antitumor activity of dosage regimens of HB-201 and HB-202 alone of in combination with pembrolizumab, using RECIST and iRECIST
Phase II Dose Expansion: Number of participants with adverse events (type, frequency, severity). | From informed consent through 30 days after last dose
  Assess the safety and tolerability of dosage regimens of HB-201 and HB-202 alone or in combination with pembrolizumab by monitoring the type, frequency, and severity of AEs and SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Development, Study Director — Hookipa Biotech GmbH
Locations (34):
- United States (26):
  - O'Neal Comprehensive Cancer Center at UAB, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arkansas for Medical Sciences, Cancer Institute, Clinical Trials Office, Fayetteville, Arkansas
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA (University of California, Los Angeles), Los Angeles, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical School, Maywood, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Fairway, Kansas
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Grossman School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Perlmutter Cancer Center at NYU Langone Hospital-Long Island, New York, New York
  - Montefiore-Einstein Center for Cancer Care, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Greenville Hospital System University Medical Center (ITOR), Greenville, South Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virgina Health System, Charlottesville, Virginia
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
- Amsterdam UMC, Locatie VUMC, Amsterdam, Netherlands
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No